CLINICAL TRIAL: NCT00137943
Title: Parents Matter!: Interventions to Promote Effective Parent-Child Communication About Sex and Sexual Risk Among African American Families
Brief Title: Parents Matter!: Interventions to Promote Effective Parent-Child Communication
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDC-NCHSTP-2834; CCU417720
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections; Sexually Transmitted Diseases; Pregnancy
Keywords: Parent-child communication; Primary prevention; sexual risk prevention; HIV
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Full Parent communication intervention
Behavioral: Brief Parent Communication Intervention
Behavioral: Control Parent Intervention

SUMMARY:
Parents Matter is a community-based project whose goal it is to develop and test an intervention designed to promote effective parent-child communication about sexuality in order to promote sexual health among adolescents.

DETAILED DESCRIPTION:
Participants in the intervention are African American parents or guardians who have children in the 4th or 5th grade that are 12 or younger. Recruitment was done through schools, housing authorities, community based organizations, and churches. Participants were randomly assigned to participate in one of three interventions delivered by community based interventionists. The enhanced sexuality communication intervention consists of five 2.5 hour sessions conducted over 5 weeks with booster sessions at 12 and 24 months post-intervention. The full sexual communication intervention focuses on general parenting skills and sexual communication skills using a variety of presentation modalities: group discussion, video, and role-plays. The brief sexual communication intervention consists of a single 2.5 hour session in which parents are provided with information on general parenting skills and sexual communication skills. Thus, this intervention seeks to provide the same information as the full sexual communication intervention but in a condensed format with little group participation. The control intervention is a single 2.5 hour session focusing on general child health issues such as diet and exercise rather than parenting and sexual communication.

ELIGIBILITY:
Inclusion Criteria:

The eligibility criteria for the parent-child dyad are as follows:

* The parent or guardian must be African-American
* The parent or guardian must be the primary caregiver for a child in 4th or 5th grade who is 12 or younger at the time of the 1st assessment.
* The parent or guardian and the child must have lived together continuously for at least the past 3 years and the child must spend most nights (5 or more) with the parent or guardian.
* The parent or guardian and the child must both speak English.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2210
Dates: Start 1999-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Percent of teens who have initiated sexual intercourse at 3 years post intervention

SECONDARY OUTCOMES:
Increase in parental knowledge at 1 year
Increase in parental skills at 1 year
Increase in parental comfort communicating at 1 year
Increase in parental confidence communicating at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rex Forehand, Ph.D., Principal Investigator — University of Vermont
Locations (3):
- United States (3):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Georgia, Athens, Georgia
  - Georgia State University, Atlanta, Georgia

REFERENCES:
- [Background] Forehand R, Gound M, Kotchick BA, Armistead L, Long N, Miller KS. Sexual intentions of black preadolescents: associations with risk and adaptive behaviors. Perspect Sex Reprod Health. 2005 Mar;37(1):13-8. doi: 10.1363/psrh.37.13.05. PMID 15888398
- [Background] Forehand, R., Miller, K.S., Armistead, L., Kitchick, B.A., & Long, N. (2004). Parents Matter! Program: An Introduction. Journal of Child and Families Studies, 13, 1-3.
- [Background] Dittus, P., Miller, K.S., Kotchick, B.A., & Forehand, R. (2004). Why parents matter: The conceptual basis for a community-based HIV prevention program prevention program for African American youth. Journal of Child and Family Studies, 13, 5-20.
- [Background] Ball, J., Pelton, J., Forehand, R., Long, N., & Wallace, S. (2004). Methodological overview of the Parents Matter! Program St. Journal of Child and Family Studies, 13, 21-34.
- [Background] Secrest, L.A., Lassiter, S.L., Armistead, L.P., Wyckoff, S.C., Johnson, J., Williams, W.B., & Kotchick, B.A. (2004). The Parents Matter! Program: Building a successful investigator community partnership. Journal of Child and Family Studies, 13, 35-45.
- [Background] Long, N., Austin, B., Gound, M., Kelly, A., Gardner, A., Dunn, R., Harris, & Miller, K. (2004). The Parents Matter! Program Interventions: Content and the facilitation process. Journal of Child and Family Studies, 13, 47-65.
- [Background] Armistead, L., Clark, H., Barber, N., Dorsey, S., Hughley, J., Favors, M., & Wycoff, S. (2004). Participant retention in the Parents Matter! Program: Strategies and outcomes. Journal of Child and Family Studies, 13, 67-80.
- [Background] Murry, V.M., Kotchick, B.A., Wallace, S., Ketchen, B., Eddings, K., Heller, L., & Collier, I. (2004). Race, culture and ethnicity: Implications for a community intervention. Journal of Child and Family Studies, 13, 81-99.
- [Background] Long, N., Miller, K.S., Jackson, L.C., Lindner, G.K., Hunt, R.G., Robinson, A.D., Goldsby, W.D., & Armistead, L.P. (2004). Lessons learned from the Parents Matter! Program. Journal of Child and Family Studies, 13, 101-112.
- [Derived] Forehand R, Armistead L, Long N, Wyckoff SC, Kotchick BA, Whitaker D, Shaffer A, Greenberg AE, Murry V, Jackson LC, Kelly A, McNair L, Dittus PJ, Lin CY, Miller KS. Efficacy of a parent-based sexual-risk prevention program for African American preadolescents: a randomized controlled trial. Arch Pediatr Adolesc Med. 2007 Dec;161(12):1123-9. doi: 10.1001/archpedi.161.12.1123. PMID 18056556